CLINICAL TRIAL: NCT05232422
Title: The Influence of Hatha Yoga Practice on Stress and Cognitive Performance
Brief Title: Yoga Practice, Stress and Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Bence Szaszkó, Principal Investigator, University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Noch fehlend
Record Dates: First submitted 2021-12-16; First posted 2022-02-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Attentional Control Switching; Task Switching Between Modalities; Inhibition; Stress; Anxiety
Keywords: anxiety; stress; mindfulness; hatha yoga; attentional control settings; attentional control theory; inhibition; shifting; task switching; cognition; attention
MeSH Terms: conditions — Inhibition, Psychological; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A pretest-posttest design is planned, with the pre- as well as the posttests each split into two sessions. Pretests are scheduled in the weeks before the intervention, posttests relatively soon after the intervention. At both data collection times, stress as well as cognitive performance (namely of attention) will be recorded in both groups (experimental group, waiting control group). While the experimental group participates in a 60-minute hatha yoga intervention at least three times a week for 8 weeks, the wait-list control group does not receive the yoga intervention until after the end of data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga-Intervention Group (Experimental): This arm will participate in a hatha yoga course for a time period of 8 weeks with a frequency of at least 3 up to 5 times per week. Further they will participate in the pre- as well as the post-tests before and after the intervention.
  Interventions: Behavioral: Hatha yoga course
- Waiting Control Group (No Intervention): For the first 8 weeks of the study this group will not receive any intervention. After the second measurement is completed they will get the possibility to participate in a hatha yoga course as well. Further they will participate in the pre- as well as the post-tests around the same time as the Yoga-Intervention group.

INTERVENTIONS:
Behavioral: Hatha yoga course — Participants will join a free hatha yoga course, conducted by a professional yoga teacher, over a time period of eight weeks with a frequency of at least three up to five times a week. The quality of the implementation of the intervention will be checked through post-monitoring by short questionnaires to be filled out by participants.
  Arms: Yoga-Intervention Group

SUMMARY:
It has been indicated in recent research that Mindfulness-based interventions may offer possibilities of promoting human stress processing and reducing anxiety or depression. They also appear to positively influence cognitive performance. One mindfulness-based intervention next to a variety of others is yoga, a combination of physical, spiritual, and mental practices of Indian origin that arose to alleviate suffering and enhance psychological and physical well-being. The goal of the study is to find out how Hatha Yoga, the most common form of yoga, consisting of stretches, yoga postures and conscious breathing, affects emotional and cognitive processes. An essential part of yoga seems to be the increase of self-regulation and consequently the regulation of stress processing and of cognitive processes in general. Building on the Attentional Control Theory, it is hypothesized that anxiety and stress limit inhibitory function - the ability to block distracting, irrelevant information - and also impair the shifting of attention that normally accompanies smooth switching between different tasks and their processing requirements. In a randomized controlled trial with an experimental and a waiting group, the investigators aim to investigate whether active participation in a 60-minute hatha yoga class (intervention) at least three times a week for two months leads to less experienced stress and improves inhibition and attentional shifting. The intervention period with pre- and postmeasurements is expected to start in early January 2022 and end in December 2022. To measure the effect of the intervention, the investigators use three experimental test tasks, one each to examine inhibition function (here, measured by distractor interference in visual search), switching between different tasks or sensory modalities (here, collected by comparing performance after passagewise alternation vs. repetition of a sound vs. light discrimination), and alternation between different stimulus features (here, determined by comparing passagewise repetition vs. alternation of target stimulus color in visual search). In all of the experimental tasks, behavioral data (reaction times and error rates) and, in two, additional electrophysiological measures (event-related potentials) are collected using EEG. To investigate the role of stress the investigators use questionnaires as well as biological stress markers from saliva. In addition, participants will receive a link to questionnaires to complete by the start of the yoga intervention. On top, trait mindfulness will be examined as a potential mechanism underlying the effects of yoga practice on attention and stress. The subjects' trait mindfulness will be assessed by questionnaire as well.

DETAILED DESCRIPTION:
Main goals of the study and hypotheses

1) What is the effect of hatha yoga on switching between tasks or sensory modalities (e.g., processing times when switching from tone to light discrimination across tasks compared to when switching from tone to light discrimination across tasks) and between features (e.g., processing times when switching from red to green target stimuli across tasks compared to when switching from red to green target stimuli across features)? The investigators hypothesize that yoga practitioners (intervention group) will show lower switching costs and lower error rates than the control group (waiting group). 2) How does hatha yoga affect the inhibition function of attention? The investigators expect increased inhibition of salient distractors (e.g., green distractors among otherwise red stimuli) during visual search (e.g., for a shape-defined target stimulus in the set of red stimuli per display) in the intervention group compared to the control group (indexed by event-related potential PD on the distractor) or lower attraction of attention by distractors (indexed by reduced N2pc on the distractor). The investigators also expect a lower rate of false alarms and a higher rate of hits in visual search performance in the intervention than in the control group. 3) What is the effect of hatha yoga on the stress and anxiety levels of the subjects? The investigators expect lower cortisol and alpha-amylase levels in the intervention group compared to the control group as well as lower levels of subjectively reported stress and reported anxiety as indicated by corresponding questionnaire scores in the intervention group compared to the control group. 4) What is the effect of Trait Mindfulness on stress parameters in the context of yoga intervention? The investigators expect that Trait Mindfulness acts as a moderator and that an increase in Trait Mindfulness during the intervention also leads to increased stress reduction.

Power analysis and recruitment strategy

Based on a power analysis with d = 0.5, 80% power and 5% alpha error, a sample size of 102 subjects is targeted, increasing to 122 with the expected dropouts of 20%. Potential participants will be made aware of the study via social media (Facebook, Instagram) and on campus via promotional materials.

Detailed description of data assessment and study materials

Interested individuals are first emailed links to screening questionnaires and given information about the study design. The investigators screen for mental disorders using mini-DIPS, a short version of DIPS (Diagnostic Interview for Mental Disorders). Individuals who meet the exclusion criteria will be excluded from the study. For those individuals who show interest in participating in the study and who do not meet the exclusion criteria (for details see "10. Eligibility"), pretest appointments will be scheduled. At the first pretest appointment, the study information will first be discussed together with the participants and written informed consent for study participation will then be obtained. The posttest appointments will run concurrently, but a consent form does not need to be signed again. In addition, the first of the three experimental cognitive tests will take place, during which behavioral measures (reaction time, error rate) will be collected in a computer experiment in the laboratory of the Faculty of Psychology.

In addition, at the first pretest/posttest appointment, participants will receive a link to the questionnaires that they must complete by the start of the yoga intervention. The self-report questionnaires include demographic data (pretest only), Perceived Stress Scale (PSS), State-Trait Anxiety Inventory (STAI)-Form Y, and Freiburg Mindfulness Inventory (FMI; long version). All mentioned questionnaires (if not specified differently) have to be completed in the pretests as well as in the posttest. In addition, the investigators use the Patient Health Questionnaire (PHQ) to characterize the sample (one-time at baseline). Questions about the feasibility of the intervention and design will be conducted using a specially constructed post-monitoring interview. As secondary outcomes, the investigators are interested in stress reactivity, which the investigators measure with the Perceived Stress Reactivity Scale (PSRS), and fatigue (Multidimensional Fatigue Inventory; MFI), as well as the control variables sleep (Pittsburgh Sleep Quality Index; PSQI), resilience (Resilience Scale RS-11), social support (Berlin Social Support Scales; BSSS), depressiveness (Beck Depression Inventory Revision; BDI- II), and self-compassion (The Self-Compassion Scale; SCS). All of these scales are assessed at pretest and at posttest. The investigators additionally assess the following data with individual items: Use of hormonal contraceptives, ongoing medication use, substance use, use of mind-body techniques, physical activity, BMI. In addition, participants receive a list of contact information for appropriate institutions to contact in the event of emergencies arising that exceed the project management's areas of expertise. At the second pretest (posttest) appointment, the investigators collect behavioral data (reaction time and error rate) as well as electrophysiological measures using EEG for the two experiments performed. Event-related potentials as well as oscillations are evaluated. In addition, independent measurement of cortisol levels and alpha-amylase will be performed on three consecutive days before and immediately after the yoga intervention - the salivary vessels for this purpose will be distributed at the first pretest appointment and the subjects will be instructed accordingly. For this, subjects will independently collect five saliva samples per day and date the exact time of collection. They will be instructed to store the samples in their own refrigerator or freezer and bring them to the Institute of Psychology before the first yoga class. Randomized assignment to experimental or control group will then occur only after the respective pretests to control for expectancy effects. If the assignment causes individuals to drop out of the study, resulting in a significant imbalance in group size, additional subjects will be recruited for the respective group.

Detailled description of the experiments

Experiment 1: Inhibition

In order to find out how the intervention also affects participants' inhibition ability, the investigators use an experimental task. The experiment consists of 36 blocks, each containing 56 trials, and 112 practice sessions. Thus, the experiment lasts approximately one hour with breaks. At the beginning of each block, subjects are presented with a target stimulus randomly selected from one of nine letters. This target stimulus can be of two different sizes (large or small). Should a run contain the target stimulus in the correct size, subjects must press the "K" key on their keyboard.

There are four different conditions: 1) trials that include a target stimulus (576 trials in total), 2) trials that include a target stimulus-like distractor, i.e., the same letter in a different size, 3) trials involving a salient distractor (a different letter in a color that is different from all other stimuli presented in the target stimulus display; 576 trials in total), 4) trials that did not meet any of the above conditions (288 trials in total).

A fixation cross is shown throughout each trial, as is usual for EEG experiments. Stimuli are presented for 200 ms, followed by a variable interstimulus interval between 800 and 900 ms. The color of the stimuli shown in the target stimulus display is randomly selected in each trial from the two possible colors, red and green, with equal probability in order to exclude color-specific effects. An exception is the salient distractor in condition 3, which is always displayed in the other color. The investigators expect different event-related potentials in the different conditions: In conditions 1) and 2) an N2pc, indicative of shifting attention, and in condition 3) a Pd, indicative of suppression of the stimulus.

Experiment 2: Task Switching

A proven method to assess the functioning of the second function affected by anxiety, the shifting function, is to use paradigms that allow for the switching between different tasks as well as between different Attention control settings. For the former, the investigators would like to use an experimental paradigm in which the investigators measure oscillations in the brain by means of EEG, which are called visually evoked steady-state potentials (SSVEP) and auditory steady-state responses (ASSR), respectively. They are measured by the Presentation of repetitive auditory and visual stimuli. It was found in past studies, that the endogenous brain oscillations take over the frequency of presentation of the respective modality. Thus, when stimuli in the auditory and visual modalities are presented with different frequencies, the investigators obtain millisecond information about which modality is currently attended. Our experiment has no distinct trials, instead stimuli are presented continuously for 180 seconds before a pause, the length of which can be determined by the subjects themselves. The trial consists of 16 blocks and the experiment lasts approximately 65 minutes with breaks.

The investigators use a 2-back task for this. Stimuli from the visual and auditory domains are presented in different frequencies and the participants have to press a key when stimulus n-2 matches stimulus n (with a stimulus gap in between). In the visual domain, a colored rectangle is presented in the center of each screen. In the auditory domain, tones with a volume of 65 dB are played one after the other.The stimuli are played simultaneously in both modalities, a distinct bimodal cue, that is played or presented in one of the modalities instead of one of the stimuli, gives an indication to which modality attention should be paid. The visual stimuli differ in color, the auditory stimuli vary in pitch. The investigators expect faster changes between the tasks in the intervention group, as well as a lower error rate.

Experiment 3: Switching between different attentional control settings

To investigate the ability to switch between stimulus features, i.e., different attentional control settings, the investigators use a contingent capture protocol. Here, the target stimuli to be responded differ in their features (such as color), which in turn results in the need for switching between the Attentional control settings. In this experiment, there are two conditions, each of which is presented in different blocks (A-B-A-B or B-A-B-A, balanced across subjects). While in one-color blocks the target stimulus is presented exclusively in the color defined at the beginning of the block, in two-color blocks there are two target colors, namely red and green, one of which always appears in the target stimulus display.

A pass proceeds as follows: First, against a black background, a fixation display is presented for a duration of 1000ms. The subsequent cueing display contains four gray rings and is shown for a duration of 50ms. Here, one of the rings takes the target color (or in two-color blocks one of the target colors) (matching cue), while the other three remain gray, or it takes on another color, namely blue (nonmatching cue). In addition, it is varied whether the cue appears at the location of the target stimulus, i.e., is valid, or not, i.e., is invalid. Following an interstimulus interval of 100 ms, the target display now appears for 150ms. In this target display, all rings get a color, but only one of them is in the target color, while two of the three remaining rings are yellow and the remaining ring with equal probability is either magenta or cyan. In addition, during the target display, all circles contain a T tilted to the left or right. The participants are asked to indicate the orientation of the T within the target color circle by pressing the right key (key y for left-tilted and m for right-tilted). In the two-color block, the color of the target stimulus changes in run n+1 compared to run n with a 50 percent probability, so the investigators get equal numbers of trials with target color repeats and target color changes and can derive switching costs from this. The investigators can also derive mixing costs from the reaction times of the different conditions (one vs. two-color block), indicative of the use of different attentional control settings. Before the task, the investigators will instruct participants to respond as quickly and accurately as possible. They will also receive written feedback on their performance by displaying "Wrong" on the PC screen for incorrect responses and "Respond Faster" for 500ms each for response times longer than 1200ms. at There will be a total of 4 blocks of 240 trials each with varying condition blocks and 24 practice trials each, resulting in an approximate duration of 75 minutes for the experiment, including breaks.

ELIGIBILITY:
Inclusion Criteria:

* healthy individual without mental or neurological disorder or disease
* 18-40 years

Exclusion Criteria:

* Insufficient comprehension of the German language
* Current mental or neurological disorders (except eating disorders)
* Current or regular yoga practice in the past
* Uncorrected visual or auditive impairment
* Scull fractures or head concussions within the last 6 weeks
* Non-existence of a vaccination or convalescence certificate of COVID-19

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Change in switching between Attentional Control Sets | Baseline plus 8 weeks
  Switching between Attentional Control Sets will be measured by switching costs, meaning longer response times (RTs) for trial-by-trial switches than repetitions of a task, and hit rate. Both variables will be combined to assess the change in ability to switch between processing different features which is expected in the intervention group in comparison to the waiting control group.
Change in task switching between modalities | Baseline plus 8 weeks
  Task switching between modalities will be measured by speed regarding switches between modalities and error rate in the respective (auditive and visual) modalities. The ability to switch between different modalities is expected to have changed in the intervention group in comparison to the waiting control group. Switching speed will be analyzed by using steady-state visual evoked potentials and auditory steady-state potentials (both measured with EEG) with tagged frequencies.
  Switching speed and error rate will be combined to report task switching ability between modalities.
Change in inhibition function | Baseline plus 8 weeks
  Inhibition function will be measured by response time, hit rate and number of false alarms.
  In addition, dependent electrophysiological variables will be the mean amplitudes of two event-related potential components, named N2-posterior contralateral (N2pc) and distractor positivity (Pd). Named variables will be combined to assess the change in inhibition function that is expected in the intervention group vs. the control group.
Change in attention shifting | Baseline plus 8 weeks
  Attention shifting will be measured by an event-related potential named N2-posterior-contralateral (N2pc) with EEG. When target-similar items are processed, N2pc should be different in the intervention group than in the control group.
Change in self-reported stress | Baseline plus 8 weeks
  Self-reported stress will be measured with the Perceived Stress Scale (PSS), ranging from 0 to 40 points, with higher scores indicating higher perceived stress.
Change in physiological stress | Baseline plus 8 weeks
  Physiological stress levels will be measured by biological markers (cortisol and alpha-amylase). Both are expected to have changed in the intervention group in comparison to the waitlisted control group, indicated by changed cortisol levels as well as changed alpha-amylase concentration.
  Both cortisol and alpha-amylase levels will be combined to report physiological stress.
Change in self-reported anxiety | Baseline plus 8 weeks
  Self-reported anxiety will be measured with the State-Trait-Anxiety Inventory (STAI) form Y, ranging from 20 to 80, with higher scores correlating with higher anxiety.
  Self-reported anxiety is expected to have changed in the intervention group in comparison to the waitlisted control group.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Ansorge, Univ.-Prof. Dr., Study Chair — University of Vienna
Locations (1):
- University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Busel C, Pomper U, Ansorge U. Capture of attention by target-similar cues during dual-color search reflects reactive control among top-down selected attentional control settings. Psychon Bull Rev. 2019 Apr;26(2):531-537. doi: 10.3758/s13423-018-1543-5. PMID 30402797
- [Background] Eysenck MW, Derakshan N, Santos R, Calvo MG. Anxiety and cognitive performance: attentional control theory. Emotion. 2007 May;7(2):336-53. doi: 10.1037/1528-3542.7.2.336. PMID 17516812
- [Background] Norcia AM, Appelbaum LG, Ales JM, Cottereau BR, Rossion B. The steady-state visual evoked potential in vision research: A review. J Vis. 2015;15(6):4. doi: 10.1167/15.6.4. PMID 26024451
- [Background] Sawaki R, Luck SJ. Capture versus suppression of attention by salient singletons: electrophysiological evidence for an automatic attend-to-me signal. Atten Percept Psychophys. 2010 Aug;72(6):1455-70. doi: 10.3758/APP.72.6.1455. PMID 20675793
- [Background] Monsell S. Task switching. Trends Cogn Sci. 2003 Mar;7(3):134-140. doi: 10.1016/s1364-6613(03)00028-7. PMID 12639695
- [Background] de Jong R, Toffanin P, Harbers M. Dynamic crossmodal links revealed by steady-state responses in auditory-visual divided attention. Int J Psychophysiol. 2010 Jan;75(1):3-15. doi: 10.1016/j.ijpsycho.2009.09.013. Epub 2009 Oct 9. PMID 19819271
- [Result] Saupe K, Schroger E, Andersen SK, Muller MM. Neural mechanisms of intermodal sustained selective attention with concurrently presented auditory and visual stimuli. Front Hum Neurosci. 2009 Nov 30;3:58. doi: 10.3389/neuro.09.058.2009. eCollection 2009. PMID 20011221
- [Derived] Szaszko B, Schmid RR, Pomper U, Maiworm M, Laiber S, Lange MJ, Tschenett H, Nater UM, Ansorge U. Testing the impact of hatha yoga on task switching: a randomized controlled trial. Front Hum Neurosci. 2024 Nov 5;18:1438017. doi: 10.3389/fnhum.2024.1438017. eCollection 2024. PMID 39568547
- [Derived] Szaszko B, Schmid RR, Pomper U, Maiworm M, Laiber S, Tschenett H, Nater UM, Ansorge U. The influence of hatha yoga on stress, anxiety, and suppression: A randomized controlled trial. Acta Psychol (Amst). 2023 Nov;241:104075. doi: 10.1016/j.actpsy.2023.104075. Epub 2023 Nov 4. PMID 37931334

DOCUMENTS (1):
  • Informed Consent Form (2021-12-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT05232422/ICF_000.pdf